CLINICAL TRIAL: NCT03860077
Title: Impact of Nicotine Reduction on Adolescent Cigarette Use, Alternative Tobacco Use, and Harm From Tobacco
Acronym: SIREN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA047356 (NIH); 1R01DA047356-01 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-03-01 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Nicotine Dependence, Cigarettes, Uncomplicated
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Very Low Nicotine Content Cigarettes (Experimental)
  Interventions: Drug: Very Low Nicotine Content Cigarettes
- Normal Nicotine Content Cigarettes (Active Comparator)
  Interventions: Drug: Normal Nicotine Content Cigarettes

INTERVENTIONS:
Drug: Very Low Nicotine Content Cigarettes — Very Low Nicotine Content Cigarettes
  Arms: Very Low Nicotine Content Cigarettes
Drug: Normal Nicotine Content Cigarettes — Normal Nicotine Content Cigarettes
  Arms: Normal Nicotine Content Cigarettes

SUMMARY:
Adolescents are an important vulnerable population to consider as the FDA moves toward a nicotine reduction policy. Such a policy, which would mandate a reduction of nicotine in all commercially available cigarettes, has the potential to transform public health and greatly reduce the toll of tobacco-related death and disease. Yet, data on the effects of such a policy on cigarette use among adolescents are lacking. Further, the advent of e-cigarettes and the popularity of alternative tobacco products have fundamentally altered the current landscape of nicotine delivery, and these products are widely used by adolescents. Although adolescent cigarette use is at an all-time low in the U.S., this reduction has been mirrored by an increase in e-cigarette use, and multiple tobacco product (MTP) use is the most common pattern of use in youth. Adolescent MTP users are more likely to be dependent on nicotine and to have begun using tobacco earlier than their single-product using peers. Thus, MTP-using youth differ from youth who solely smoke cigarettes in meaningful ways that have implications for responses to a nicotine reduction regulatory policy. In adults, longer-term studies have demonstrated that very low nicotine content (VLNC) cigarette exposure results in fewer cigarettes smoked and reduced toxicant exposure; however, increased use of alternative tobacco products has also been reported. No studies to date have examined the effects of VLNC cigarettes on MTP use or toxicant exposure in youth. This study will use real-time, smartphone-based ecological momentary assessment (EMA) and laboratory-based assessments to: (1) investigate the effects of cigarette nicotine reduction on cigarette and MTP use, (2) assess the influence of cigarette nicotine reduction on the harms associated with tobacco use, including nicotine and toxicant exposure, respiratory symptoms, perceived health risk and nicotine dependence, and (3) use a combination of laboratory and real-time assessment to investigate the effects of nicotine reduction on changes in withdrawal, craving, and the reinforcing efficacy of cigarettes to characterize the mechanisms by which VLNC use may affect behavior. Overall, this project will help determine the effects of VLNC cigarettes on real-world tobacco use behavior and indices of tobacco-related harm in adolescents, and examining the mechanisms through which nicotine reduction in cigarettes may effect such changes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Ages 15-20 inclusive 2) Male and female current daily smokers

  1. Defined as self-reported daily cigarette smoking at phone screening AND
  2. a breath carbon monoxide (CO) criterion of 5 ppm or higher; if this is not met, urine cotinine levels, detected by a NicAlert cotinine screening device, must indicate recent smoking (level 3 or higher) 3) Current users of alternative tobacco product(s)

  a. Defined as any self-reported use of at least one non-cigarette tobacco product (e.g., e-cigarettes, little cigars, cigarillos, hookah, etc.) in the past 30 days 4) Participants must speak and comprehend English well enough to complete study procedures.

  a. Participant will be asked to read aloud first few lines of informed consent and then summarize the contents aloud to check for competency 5) Participants under 18 must provide assent and parental consent from a parent/guardian.

  a. Participants age 18 or 19 may provide their own written consent contingent on photo ID verification of age.

Exclusion Criteria:

* 1) Unwilling to use research cigarettes as part of the study 2) Self-reported daily drinking of alcohol or use of illicit or non-prescribed drugs (excluding marijuana) > 10 days in the past 30 days

  a. We will ask about daily alcohol and drug use in the phone screen, and we will use the Timeline Follow-Back to assess current and recent marijuana and alcohol use.

  3) Currently seeking treatment to quit smoking, and/or intending to quit smoking for good in the next 30 days
  1. This information corresponds to questions 2 & 3 of the Stages of Change measure which will be administered at the in-person screening.
  2. These participants will be excluded, and provided with referral information for cessation services in the community.

     4) Suicidal ideation in the past month or any past-year suicide attempts

  a. Suicidal ideation determined by the MINI ( Mini International Neuropsychiatric Interview) suicide subscale at the in-person screening (Questions 4 and 5) b. Suicide attempt in the past year determined by MINI question 6.a. (If participant has a lifetime history of suicide attempt between 1 and 10 years ago, licensed medical monitor approval required) c. If a participant indicates that he/she currently has suicidal ideation during this or any future session, the Emergency Protocol will be followed in which a Licensed Clinician will be contacted immediately, and participants will speak with the clinician over the phone and the clinician will determine the appropriate action to take to keep the child safe.

  5) Pregnant or breastfeeding

  a. Determined by urine test at in-person screening; tested again at each in-person visit; participant will be excluded or withdrawn if test indicates pregnancy b. Self-reports current breastfeeding at in-person screening 6) Any medical or psychiatric conditions in which participation is likely to pose a significant threat to health or for which the condition could interfere with the ability of the participant to fully participate (as determined by LMP).

  7) Having participated in another research study during the past year in which they were switched to research cigarettes for longer than one week.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Cassidy, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators involved in this project intend to share findings from its research through publications and presentations. After all data have been collected and the results of the study have been published, de-identified data will be made available to other qualified investigators upon request. Institutions and/or individuals wishing to access any resources or data must contact the Principal Investigators. Persons requesting data must do so in writing, identifying their affiliation and how and by whom the data will be used. The request will be evaluated by the PIs and Co-Investigators to ensure that it meets reasonable demands of scientific integrity.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were consented at Screening/Baseline 1 (N=57). Those who remained eligible and interested were randomized at Baseline 2 (N=49). Participant flow was documented for randomized participants.
Groups:
- Normal Nicotine Content Cigarettes: Normal Nicotine Content Cigarettes:15.8 mg/g nicotine per cigarette
- Very Low Nicotine Content Cigarettes: Very Low Nicotine Content Cigarettes: 0.4 mg/g nicotine per cigarette
Period: Overall Study
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Started | 25 | 24
Completed | 21 | 17
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Population: Characteristics of randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.72 (0.73) | 19.08 (0.88) | 18.90 (0.82)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 13 | 9 | 22
  Female | 8 | 13 | 21
  Transgender, genderqueer, or other identity not listed | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 17 | 32
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes smoked per day] | 6.3 (4.4) | 7.6 (7.4) | 6.9 (6.0)
Carbon Monoxide [Mean (Standard Deviation); unit: parts per million] — Exhaled breath carbon monoxide
  parts per million | 10.4 (9.6) | 11.5 (11.7) | 11.02 (10.6)
Baseline Number of Other Tobacco Use Days in Past 30 [Mean (Standard Deviation); unit: Days in past 30 days] | 4.32 (5.70) | 5.7 (3.5) | 5.0 (3.61)

OUTCOME MEASURES:

1. Primary Outcome: Average Cigarettes Smoked Per Day
Description: Average number of cigarettes (study and non-study) smoked in the past week prior to the final session.
Time Frame: Week 4
Population: Participants who completed week 4
Measure: Mean (Standard Deviation); unit: average cigarettes per day
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 21 | 17
average cigarettes per day | 4.3 (2.6) | 8.0 (10.33)
Statistical Analysis 1: Comparison: Normal Nicotine Content Cigarettes vs Very Low Nicotine Content Cigarettes; These are results of a 2-group (VLNC & NNC) x 2 repeated measures (Baseline & Week 4) mixed effects model to test the effect of the randomization group (VLNC vs. NNC) on change in cigarette use and alternative tobacco product (ATP) use from Baseline to Week 4. Group (VLNC vs. NNC) is a fixed, between-subjects focal predictor. Timepoint (Baseline vs. Week 4) is a fixed, within-subjects repeated measure. Subject is a random effect, accounting for variability in Baseline cigarette and ATP use; Test type: Superiority — Average cigarettes per day was positively skewed, with a non-normal residual distribution in a mixed model analysis specifying a normal (Gaussian) outcome distribution. Therefore, this outcome was recoded to integers and modeled as a count with a negative binomial distribution and log link. The focal test is the difference in change from Baseline to Week 4 (i.e., Time) in the VLNC vs. NNC condition (i.e., Group), which is a cross-level interactive effect of Time and Group; p = .111, Mixed Models Analysis; Risk Ratio (RR) = 1.42, 95% CI 2-sided [0.92 to 2.19], Standard Error of Mean 0.21 — The reported value is the standard error of the mean for the non-exponentiated estimate = 0.35

2. Primary Outcome: Average Number of Days of Combustible and Noncombustible Use
Description: Average number of days of combustible and noncombustible use. This measure is a sum of the days of combustible use (out of 7 days) and noncombustible use (out of 7 days) recorded in the week prior to week 4, averaged over 14 days. As this measure is a sum of the two variables, its possible range is 0-14.
Time Frame: Week 4
Population: Those who completed Week 4 are included in the outcome means.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 21 | 17
days | 4.80 (3.12) | 5.17 (3.87)
Statistical Analysis 1: Comparison: Normal Nicotine Content Cigarettes vs Very Low Nicotine Content Cigarettes; This outcome was recoded as a dichotomous outcome with a binary distribution and log link. The focal test is the difference in change from Baseline to Week 4 (i.e., Time) in the VLNC vs. NNC condition (i.e., Group), which is a cross-level interactive effect of Time and Group; Test type: Superiority; p = .721, Mixed Models Analysis; Odds Ratio (OR) = .71, 95% CI 2-sided [.11 to 4.75], Standard Error of Mean .93 — The reported value is the standard error of the mean for the non-exponentiated estimate = - 0.34

3. Secondary Outcome: Amount of Noncombustible Alternative Product Use
Description: Number of days of noncombustible tobacco product use in the past 7 days prior to week 4
Time Frame: Week 4
Population: Those who completed week 4.
Measure: Mean (Standard Deviation); unit: average days
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 21 | 17
average days | 4.76 (3.11) | 4.29 (3.4)
Statistical Analysis 1: Comparison: Normal Nicotine Content Cigarettes vs Very Low Nicotine Content Cigarettes; Test type: Superiority — Frequencies of non-combustible alternative product use (ATP) were bimodal with peaks at 0 (no use) and 7 (daily use). Therefore, this outcome was recoded as a dichotomous outcome with a binary distribution and log link. The focal test is the difference in change from Baseline to Week 4 (i.e., Time) in the VLNC vs. NNC condition (i.e., Group), which is a cross-level interactive effect of Time and Group; p = .564, Mixed Models Analysis; Odds Ratio (OR) = .57, 95% CI 2-sided [.08 to 3.99], Standard Error of Mean 0.96 — The reported value is the standard error of the mean for the non-exponentiated estimate = - 0.56

4. Secondary Outcome: Average Study Cigarettes Per Day
Description: Average number of study cigarettes smoked per day across 7 days prior to week 4
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: average cigarettes per day
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 21 | 17
average cigarettes per day | 3.32 (2.86) | 4.98 (5.92)
Statistical Analysis 1: Comparison: Normal Nicotine Content Cigarettes vs Very Low Nicotine Content Cigarettes; The study cigarette outcome is modeled with a normal, Gaussian distribution. The focal test is the difference in change from Baseline to Week 4 (i.e., Time) in the VLNC vs. NNC condition (i.e., Group), which is a cross-level interactive effect of Time and Group. Baseline in this analysis is average number of usual brand cigarettes at baseline, prior to randomization; Test type: Superiority; p = .876, Mixed Models Analysis; Slope = .25, 95% CI 2-sided [-2.92 to 3.42], Standard Error of Mean 1.56

5. Secondary Outcome: Toxicant Exposure
Description: Total Nicotine Equivalents (TNEs)
Time Frame: Week 4
Population: All participants who provided urine data at Week 4, and for whom there were analyzable levels of TNEs.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 19 | 15
ng/ml | 3875.395 (4700.761) | 6284.507 (6641.2956)
Statistical Analysis 1: Comparison: Normal Nicotine Content Cigarettes vs Very Low Nicotine Content Cigarettes; Test type: Superiority — The focal test is the difference in change from Baseline to Week 4 (i.e., Time) in the VLNC vs. NNC condition (i.e., Group), which is a cross-level interactive effect of Time and Group; p = .226, Mixed Models Analysis; Slope = -2166.79, 95% CI 2-sided [-5743.04 to 1409.47], Standard Error of Mean 1753.48

6. Other Pre Specified Outcome: American Thoracic Society Questionnaire
Description: Respiratory Health Symptoms; an 8-item questionnaire measuring frequency of experience respiratory symptoms; scores can range from 8 to 40 and greater scores indicate greater frequency.
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Perceived Health Risk Questionnaire
Description: Perceived risk for developing diseases associated with use study cigarettes and usual brand cigarettes; Scores range from 1 (much less risk) to 5 (much greater risk) for each disease
Time Frame: Week 4
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Nicotine Dependence
Description: Modified Fagerstrom Tolerance Questionnaire (mFTQ) score; Scale 2-8, higher scores indicate greater nicotine dependence
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Craving
Description: Questionnaire on Smoking Urges (QSU) post- smoking in the laboratory, a 10 item scale that is comprised of 2 factors; Factor 1 included items 1, 3, 6, 7, and 10 Factor 2 included items 2, 4, 5, 8, and 9 The score for each factor is calculated by summing the item scores; the total score is calculated by summing all 10 items. A single-item craving question (ranging from 1-10, not all to greatly) from daily random and post-event Ecological Momentary Assessments.
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Withdrawal
Description: Minnesota Nicotine Withdrawal Scale 7-item version; greater score indicates greater withdrawal
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Subjective Response to Cigarettes
Description: Cigarette Evaluation Scale post-smoking in the laboratory; 5 subscales are derived from this scale: Psychological Reward, Smoking Satisfaction, Enjoyment of Respiratory Sensations, Craving Reduction; Aversion. Event level on satisfaction derived from post-use responses on daily Ecological Momentary Assessments.
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Hypothetical Purchasing of Cigarettes
Description: Cigarette Purchase Task; Five indices of demand for cigarettes are derived from this measure (Intensity, Omax, Breakpoint, Pmax, Alpha)
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Hypothetical Purchasing of Tobacco Products
Description: Purchasing of cigarettes and other tobacco products across changing prices in Experimental Tobacco Marketplace task
Time Frame: Baseline-Week 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

LIMITATIONS AND CAVEATS:
The study enrollment was slowed due to programming of the smartphone app; we intended to make up enrollment numbers, however, the COVID-19 pandemic severely affected our ability to recruit. We lost several months of recruitment due to shutdowns, and post-COVID recruitment rates were much lower than pre-COVID; perhaps due to concerns about in-person sessions despite measures taken to reduce contact.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (5):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03860077/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03860077/SAP_001.pdf
  • Informed Consent Form: 18+ Consent (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03860077/ICF_002.pdf
  • Informed Consent Form: Parental Consent Form (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03860077/ICF_003.pdf
  • Informed Consent Form: Minor Assent Form (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03860077/ICF_004.pdf